CLINICAL TRIAL: NCT00116493
Title: Evaluation of Anthelminthics and Multivitamins for Treatment of Severe Anemia in Pregnant Women and Children 6-24 Months of Age in Pakistan
Brief Title: Severe Anemia Treatment Trials, Pakistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Parul Christian, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: H.22.03.04.22.A2; Thrasher Research Fund 02817-9
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Anemia
Keywords: severe anemia; anthelminthic; multivitamins; pregnancy; children; Pakistan
MeSH Terms: conditions — Anemia | interventions — Mebendazole; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Standard of care (Iron-folic acid + Deworming)
  Interventions: Dietary Supplement: Iron-folic acid and mebendazole
- 2 (Experimental)
  Interventions: Drug: Mebendazole
- 3 (Experimental)
  Interventions: Dietary Supplement: Multivitamins
- 4 (Experimental)
  Interventions: Drug: Mebendazole + Multivitamin

INTERVENTIONS:
Dietary Supplement: Iron-folic acid and mebendazole — 100 mg iron for pregnant women, 25 mg iron for children
  1 mg of folic acid for pregnant women, 100 ug folic acid for children 500 mg of mebendazole for both pregnant women and children
  Arms: 1
Drug: Mebendazole — 100 mg twice a day for 3 days; Iron-folic acid also given
  Arms: 2
Dietary Supplement: Multivitamins — Iron-folic acid also given; Includes vitamins A, C, B12, E, and B2
  Arms: 3
Drug: Mebendazole + Multivitamin — Multivitamins + Mebendazole at 100 mg twice a day for 3 days; Iron-folic acid also given
  Arms: 4

SUMMARY:
The purpose of this study is to test the efficacy of two enhanced regimens (deworming and multivitamins) in the treatment of severe anemia in pregnant women and children 6-24 months of age in Karachi, Pakistan.

DETAILED DESCRIPTION:
Anemia continues to be a public health problem of global proportions. Severe anemia (hemoglobin, Hb< 70 g/L) is of special concern as it poses a significant health and mortality risk. Pregnant women and young children (6-24 months of age) are the two groups at highest risk. Severe anemia in pregnant women is associated with an elevated risk of maternal and perinatal mortality as well as case fatality. Pakistan, the country in which this study is ongoing, may harbor the highest prevalence of severe anemia in South Asia, with as high as 15% being reported among pregnant women. Comparable rates (11-12%) are also seen among 6-24 month old children. Iron deficiency is one of the major causes of anemia in young children and pregnant women in South Asia. In addition to iron, deficiency of vitamins such as folic acid, vitamin A, vitamin C, riboflavin and vitamin E can also inhibit erythropoiesis. Apart from these nutritional causes, two other infectious causes of severe anemia are malaria and geohelminths. The current international recommendation for treatment of anemia includes iron and folic acid but not other vitamins.

Comparisons: Severely anemic pregnant women and children 6-24 months are randomized to receive enhanced treatment of deworming and multivitamins over and above the standard of care of iron-folic acid using a 2x2 factorial design.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with severe anemia (Hb<70g/L)
* Children 6-24 months with severe anemia (Hb<70 g/L)

Exclusion Criteria:

* Gestational age >=36 weeks
* Edema
* Breathlessness

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1009 (Actual)
Dates: Start 2004-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Severe Anemia

CONTACTS AND LOCATIONS:
Overall Officials: Parul Christian, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Bhutta Z, Klemm R, Shahid F, Rizvi A, Rah JH, Christian P. Treatment response to iron and folic acid alone is the same as with multivitamins and/or anthelminthics in severely anemic 6- to 24-month-old children. J Nutr. 2009 Aug;139(8):1568-74. doi: 10.3945/jn.108.103507. Epub 2009 Jun 17. PMID 19535425
- [Result] Christian P, Shahid F, Rizvi A, Klemm RD, Bhutta ZA. Treatment response to standard of care for severe anemia in pregnant women and effect of multivitamins and enhanced anthelminthics. Am J Clin Nutr. 2009 Mar;89(3):853-61. doi: 10.3945/ajcn.2008.26826. Epub 2009 Jan 28. PMID 19176737